CLINICAL TRIAL: NCT01251198
Title: Stent For Life Observatory
Acronym: SFL
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Principal Investigator, Martine Gilard, Professor, French Cardiology Society
Other Study IDs: Stent For Life
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute coronary Syndrome: Patients affected are patients with acute coronary syndrome with ST segment elevation ST (myocardial infarction) in 48 hospitalized in one of the centers (emergency, ambulance, intensive care unit, cardiac catheterization lab).

SUMMARY:
Observatory multicenter, prospective, to support the acute phase of acute coronary syndromes with ST segment elevation ST (myocardial infarction).

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a myocardial infarction less than 48 hours during the November 2010 is eligible and should be considered for inclusion in the study.
* Every patient who agreed to participate in the study

Exclusion Criteria:

* Patients with myocardial infarction after a coronary revascularization, or after cardiac surgery or extra heartbeat.
* Patient denying that his personal data are subject to treatment automated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected are patients with acute coronary syndrome with ST segment elevation ST (myocardial infarction) in 48 hospitalized in one of the centers (emergency, ambulance, intensive care unit, cardiac catheterization lab).
Sampling Method: Non-Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martine Gilard, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CHU Brest, Brest, France

REFERENCES:
- [Background] Cambou JP, Simon T, Mulak G, Bataille V, Danchin N. The French registry of Acute ST elevation or non-ST-elevation Myocardial Infarction (FAST-MI): study design and baseline characteristics. Arch Mal Coeur Vaiss. 2007 Jun-Jul;100(6-7):524-34. PMID 17893635
- [Background] Simon T, Verstuyft C, Mary-Krause M, Quteineh L, Drouet E, Meneveau N, Steg PG, Ferrieres J, Danchin N, Becquemont L; French Registry of Acute ST-Elevation and Non-ST-Elevation Myocardial Infarction (FAST-MI) Investigators. Genetic determinants of response to clopidogrel and cardiovascular events. N Engl J Med. 2009 Jan 22;360(4):363-75. doi: 10.1056/NEJMoa0808227. Epub 2008 Dec 22. PMID 19106083